CLINICAL TRIAL: NCT01722864
Title: An Open Label Safety Study of COV155 in Subjects With Osteoarthritis or Chronic Low Back Pain
Brief Title: Open Label Safety and Tolerability Study of COV155 in Subjects With Osteoarthritis (OA) or Chronic Low Back Pain (CLBP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COV15010233
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Chronic Low Back Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COV155 (Experimental): COV155, loading dose of 3 tablets followed by 2 tablets every 12 hours for 10 to 35 days.
  Interventions: Drug: COV155

INTERVENTIONS:
Drug: COV155 — COV155 tablets
  Other Names: MNK155

SUMMARY:
A study to show the safety of COV155 in patients with osteoarthritis of the knee or hip or moderate to severe chronic low back pain.

ELIGIBILITY:
Inclusion Criteria

* General good health, other than osteoarthritis (OA) or chronic low back pain (CLBP), based upon results of medical and surgical history and medical exam
* ≥18 years of age
* Voluntarily provide written informed consent
* Female subjects eligible if

  1. Not pregnant or lactating; not planning to become pregnant within next 60 days
  2. Surgically sterile, or 2 years postmenopausal, or practicing acceptable birth control for more than 60 days prior to Screening and use of acceptable birth control during the study and 7 days following the last dose of COV155
* Male subjects biologically capable of having children must use reliable birth control during study and 7 days after the last dose of COV155. Surgical sterilization of the subject's monogamous partner qualifies as adequate birth control
* Clinical diagnosis of one of the following

  1. OA of knee or hip for at least 1 year with moderate to severe daily pain despite chronic use of stable doses of non-steroidal anti-inflammatory drugs (NSAIDs) or other non-steroidal, non-opioid therapies or with therapy including opioids
  2. Moderate to severe CLBP for at least several hours a day for a minimum of 90 days, not due to a known malignancy, and classified as non-neuropathic, neuropathic, or symptomatic for more than 6 months after LBP surgery
  3. OA of knee and scheduled to undergo unilateral primary tricompartmental arthroplasty.
* For CLBP/OA: Average in-clinic pain score of ≥3 on 11-point (0 to 10) numerical rating scale (NRS) as an average for the last 24 hours at Screening; - Pain intensity score of ≥4 on NRS as an average for the last 24 hours at Baseline
* For TKR: 11. Post-operative pain intensity scores ≥ 4 on a 0 to 10 NRS after discontinuation of post-surgical patient controlled analgesia or intravenous pain medications; body mass index ≤ 38.0; classified as either Physical Status (PS)-1 or PS-2.

Exclusion Criteria

* Any clinically significant condition or unstable illness that precludes study participation or interferes with assessment of pain and other symptoms of CLBP or OA or would increase the risk of opioid or NSAID related adverse events
* Schizophrenia or an uncontrolled or poorly controlled major psychiatric condition or clinically significant anxiety or depression
* Active malignancy or history of malignancy within 2 years prior to Screening other than dermal or cervical squamous cell carcinoma in situ
* History of seizures (exception-pediatric febrile seizures)
* Clinically significant ECG abnormalities or uncontrolled hypo- or hypertension
* For CLBP/OA: Arthroscopic or open surgery on either the knee or hip selected as primary OA study joint within 6 months prior to Screening; - For CLBP subjects, a surgical procedure for back pain within 6 months prior to Screening, nerve or plexus block within 30 days prior to Screening or botulinum toxin injection in lower back region within 90 days prior to Screening. For OA subjects, joint injection within 30 days prior to Screening; - Surgical implants of either the knee or hip selected as the primary OA joint; history of spinal stenosis (only CLBP subjects)
* For TKR: Major prior open knee surgery on same side as arthroplasty; any other surgery/elective procedures within 4 weeks of Screening, or during study; going to rehabilitation after surgery
* Gastric reduction or gastric band surgery
* Taking opioids in equivalents to more than 20 mg hydrocodone or more than 40 mg morphine orally per day, or taking opioid medications 4 days a week or more
* Known allergy or hypersensitivity to opioids, acetaminophen or ibuprofen
* Certain lab abnormalities
* Unable to discontinue use of prohibited medications or history of substance or alcohol abuse within 2 years prior to Screening or positive urine drug test at Screening for alcohol, illicit drugs (including medical cannabis) or controlled substances other than prescribed medications
* Positive for human immunodeficiency virus, hepatitis B (surface antigen), and/or hepatitis C
* Any other chronic pain condition other than CLBP or OA that would interfere with the assessment of CLBP or OA
* Used a monoamine oxidase inhibitor, antipsychotic, or benzodiazepine within 14 days prior to Screening or started or changed doses of anticonvulsants, selective serotonin reuptake inhibitors, serotonin norepinephrine reuptake inhibitors, or tricyclic antidepressants within 30 days prior to Screening
* Previously received COV155 in a study
* Received any investigational drugs or devices within 30 days prior to Screening
* Other criteria as specified in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of COV155 | Up to 35 days
  Safety evaluations using physical exam, vital signs, clinical laboratory tests, pulse oximetry, and adverse events.

SECONDARY OUTCOMES:
Modified Brief Pain Inventory short form (mBPI-sf) - intensity | Baseline, Weeks 1, 2, 3, 4, and 5
  The mean changes from pre-treatment in the worst, least, average, and current pain using the worst, least, average, and current pain intensity items of the mBPI-sf (questions 1 to 4).
Modified Brief Pain Inventory short form (mBPI-sf) - pain relief | Baseline, Weeks 1, 2, 3, 4, and 5
  Evaluate pain relief using the pain relief item of the mBPI-sf (question 5).
Modified Brief Pain Inventory short form (mBPI-sf) - pain interference | Baseline, Weeks 1, 2, 3, 4, and 5
  Evaluate the pain-related quality of life using the Pain Interference subscale of the mBPI-sf.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Baseline, Weeks 1, 2, 3, 4, and 5
  The mean changes from pre-treatment in disease-specific quality of life using the WOMAC (48-hour version) for subjects with OA of the hip or knee.
Roland Morris/Disability Questionnaire | Baseline, Weeks 1, 2, 3, 4, and 5
  The mean changes from pre-treatment in disease-specific quality of life using the Roland Morris LBP and Disability Questionnaire for subjects with CLBP.

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Anaheim Clinical Trials, Anaheim, California
  - Orange County Research Institute, Anaheim, California
  - United Clinical Research Center, Inc., Anaheim, California
  - Torrance Clinical Research Inc., Lomita, California
  - Probe Clinical Research Corporation - Santa Ana, Santa Ana, California
  - Lake Internal Medicine Associates, Eustis, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Eastern Research, Hialeah, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Clinical Neuroscience Solutions Inc., Orlando, Florida
  - Compass Research, LLC, Orlando, Florida
  - Martin E. Hale, MD PA (Gold Coast Research LLC), Plantation, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - International Clinical Research, LLC, Sanford, Florida
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Goldpoint Clinical Research, Indianapolis, Indiana
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Independent Clinical Researchers, Las Vegas, Nevada
  - Clinical Study Center of Asheville, LLC, Asheville, North Carolina
  - Wake Research Associates LLC, Raleigh, North Carolina
  - The Center for Clinical Research LLC, Winston-Salem, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Hightop Physicians Inc./Medical Research Center, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Community Research - Anderson, Cincinnati, Ohio
  - Health Research Institute, Oklahoma City, Oklahoma
  - DeGarmo Institute for Medical Research, Greer, South Carolina
  - Pain Specialists of Charleston, North Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - FutureSearch Trials of Neurology, LP, Austin, Texas
  - Clinical Trial Network, Houston, Texas
  - ClinRx Research LLC, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia

REFERENCES:
- [Derived] Zheng Y, Kostenbader K, Barrett T, Hisaw E, Giuliani MJ, Chen Y, Young JL. Tolerability of Biphasic-Release Hydrocodone Bitartrate/Acetaminophen Tablets (MNK-155): A Phase III, Multicenter, Open-Label Study in Patients With Osteoarthritis or Chronic Low Back Pain. Clin Ther. 2015 Jun 1;37(6):1235-47. doi: 10.1016/j.clinthera.2015.03.019. Epub 2015 Apr 23. PMID 25913923